CLINICAL TRIAL: NCT04900337
Title: A Phase 1/2 Prospective Randomized Placebo Controlled Study to Assess the Safety, Tolerability and Efficacy of Amorphous Calcium Carbonate (ACC) Administered Sublingual and in Inhalation Concomitantly With BAT (Best Available Care) as Compared to Placebo and BAT for the Treatment of Moderate to Severe COVID-19 Patients.
Brief Title: Safety, Tolerability and Efficacy of Amorphous Calcium Carbonate (ACC) Compared to Placebo and Best Available Care (BAT), for the Treatment of Moderate to Severe COVID-19 Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMCS-COVID-001
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMOR 18 Powder & Inhalation (Experimental): AMOR_inhaled Double Pack- Each kit contains two tubes that after mixing result with 1.14 % ACC in 10 ml suspension.
  AMOR_powder- ACC in a dry powder (up to 2000mg Calcium/day sublingually).
  Interventions: Drug: AMOR 18 Powder & Inhalation
- Placebo (Placebo Comparator): Placebo_Inhaled Double Pack - Each kit contains two tubes of saline at different volumes (similar to investigational product) after mixing the results remains saline at a final volume of 10ml.
  Placebo_Powder: Each sachet contains powder at the same particle size and weight as the powder of the investigational product.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMOR 18 Powder & Inhalation — AMOR Inhalation x 3 times a day, via Circulaire® II AMOR Powder x 4 times a day, sublingual
  Arms: AMOR 18 Powder & Inhalation
Drug: Placebo — Placebo Inhalation x 3 times a day, via Circulaire® II Placebo Powder x 4 times a day, sublingual
  Arms: Placebo

SUMMARY:
This is a phase I/II study with Amorphous Calcium Carbonate (ACC) administered sublingual and in Inhalation concomitantly with BAT (Best Available Care) as Compared to Placebo and BAT for the treatment of Moderate to Severe COVID-19 patients. The purpose of this study is to assess the Safety, Tolerability and Efficacy of Amorphous Calcium Carbonate (ACC).

DETAILED DESCRIPTION:
This study includes two parts:

Part 1 - A training period of a single arm active treatment open label, to assess the optimal method of study drug administration, as well as the safety of the combined administration, on 5 patients.

Following DSMB review of the data collected in part 1 and the DSMB approval to proceed to next part, part 2 will be initiated.

Part 2 - A randomized (1:1) placebo controlled 2 arms study. Additional 95 patients will be recruited to this arm.

Patients who are hospitalized due to moderate or severe COVID-19 will be recruited to this study.

The following elements are the main elements that will be assessed:

1. Confirmation SARS-CoV-2 infection
2. Respiratory Function (breathing rate, SpO2 Oxygen Saturation
3. Vital Signs (BP, HR), Temperature
4. Blood Tests
5. Disease Severity Scale (8 points ordinal scale)

The whole study period per patient will be 22 days (21 treatment days) or until the patient has recovered and/or is discharged from the hospital, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of age ≥ 18 years and ≤ 80 years
2. Signed an Informed Consent
3. Agree to undergo blood tests as per protocol
4. Diagnosed with COVID-19
5. Evidence of lung involvement (by chest X rays or lung US)
6. May or may not need for Supplemental Oxygen at enrollment
7. Hospitalized

Exclusion Criteria:

1. Pregnant or breast-feeding females
2. Patients with non-COVID19 related Pneumonia
3. Any pulmonary disease not related to COVID19
4. Tracheostomy
5. High flow oxygen or non-invasive ventilation (Bipap) or Mechanical ventilation
6. Hypercalcemia defined as calcium or corrected calcium > 10.5mg/dL
7. Hyperphosphatemia defined as > 4.5mg/dL
8. Urine calcium to creatinine ratio >0.14
9. Participating in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Severity rating of Disease using an 8-point ordinal scale on days 7, 14, 21, measured as improvement greater than or equal to 1 point from baseline score. | Treatment Day 1 to Day 21 or discharge from hospital, the earliest.
  Ordinal 8 points scale:
  1. Not hospitalized and no limitations of activities.
  2. Not hospitalized, with limitation of activities, home oxygen requirement, or both.
  3. Hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infection-control or other nonmedical reasons).
  4. Hospitalized, not requiring supplemental oxygen but requiring ongoing medical care (related to Covid-19 or to other medical conditions).
  5. Hospitalized, requiring any supplemental oxygen.
  6. Hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices.
  7. Hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  8. Death.

SECONDARY OUTCOMES:
Duration of Hospital stay | Date of hospitalization to treatment day 21 or discharge, whichever comes first.
  Time to discharge from hospital
Duration of ICU stay | Treatment Day 1 to treatment day 21 or discharge, whichever comes first.
  Time patient is hospitalized in ICU, if applicable.
Duration of Mechanical Ventilation Use | Treatment Day 1 to treatment day 21 or discharge, whichever comes first.
  Time the patient requires Mechanical Ventilation (if needed)
Duration of Oxygen Supplementation | Treatment Day 1 to treatment day 21 or discharge, whichever comes first.
  Time the patient requires Oxygen Supplementation (if needed)
Duration of No Oxygen use | Treatment Day 1 to treatment day 21 or discharge, whichever comes first.
  Time the patient does not require Oxygen Supplementation
% of patients to meet ordinal scale of 3 or less | Treatment Day 1 to treatment day 21 or discharge, whichever comes first.
  Proportion of subjects hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infection-control or other nonmedical reasons).
% of death | Treatment Day 1 to treatment day 21 or discharge, whichever comes first.
  Proportion of subjects died during the study, if any.
Frequency and severity of adverse events | Screening to End of treatment day 21 or discharge, whichever comes first.
Number and percent of patients with hypercalcemia | Treatment days 4, 7, 11, 17 and 21.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Shamir MC, Be’er Ya‘aqov
  - Ziv MC, Safed
  - Tel-Aviv Sourasky MC, Tel Aviv